CLINICAL TRIAL: NCT05674305
Title: A Multicenter, Randomized, Non-inferior Phase III Study of Radiotherapy Alone Versus Concurrent Chemo-radiotherapy in Locally Advanced Nasopharyngeal Carcinoma Patients With Complete Remission of EBV DNA After One Cycle GP Regime Neoadjuvant Chemotherapy
Brief Title: Radiotherapy Alone Versus Concurrent Chemo-radiotherapy for Nasopharyngeal Carcincoma Patients With Undectable EBV DNA After One Cylce Neoadjuvant Chemotherpy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Chaosu Hu, MD and PhD, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20122229-15
Record Dates: First submitted 2022-12-30; First posted 2023-01-06 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiotherapy; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy alone (Experimental): Patients with undectable plazma EBV DNA after first cycle neoadjuvant chemotherapy using GP regimen (gemcitabine 1000mg/m2 d1,8+ cisplatin 25mg/m2 d1-3) and without rebound during the course of second and third cycle received definitive radiotherapy to head and neck region.
  Interventions: Drug: Radiotherapy
- Concurrent chemoradiotherapy (Active Comparator): Patients with undectable plazma EBV DNA after first cycle neoadjuvant chemotherapy using GP regimen (gemcitabine 1000mg/m2 d1,8+ cisplatin 25mg/m2 d1-3) and without rebound during the course of second and third cycle received definitive radiotherapy to head and neck region plus two cycles of concurent chemotherapy （cisplatin 80mg/m2）
  Interventions: Drug: Radiotherapy; Drug: Cisplatin

INTERVENTIONS:
Drug: Radiotherapy — IMRT for primary and regional field
Drug: Cisplatin — Cisplatin 80mg/m2, 21days/cycle, 2 cycles
  Arms: Concurrent chemoradiotherapy

SUMMARY:
The goal of this multicenter randomized non-inferior study is to compare radiotherapy alone versus concurrent chemoradiotherapy in locally advanced nasopharyngeal carcinoma patients whose EBV DNA drop to undetectable level after one cycle neoadjuvant chemotherapy using GP regimen. The main question it aims to answer is: the omission of concurrent chemotherapy is safe in the relatively good prognostic patients identified by the response of EBV DNA. Participants will be randomized to either radiotherapy alone or the standard treatment concurrent chemoradiotherapy if their EBV DNA decrease to undetectable level post first cycle of neoadjuvant chemotherapy and don't rebound in the second and third cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with newly histologically confirmed non-keratinizing nasopharyngeal carcinoma, type of WHO II or III.
2. Age 18-70 years.
3. Clinical stage III-IVa (based on the 8th American Joint Committee on Cancer[AJCC] edition).
4. Patients with detectable pre-treatment plasma EBV DNA but undetectable EBV DNA after one cycle neoadjuvant and no EBV DNA rebound during the second and third cycle.
5. ECOG (Eastern Cooperative Oncology Group) score: 0-1
6. Hemoglobin (HGB) ≥90 g/L, white blood cell (WBC) ≥4×109 /L, platelet (PLT) ≥100×109 /L.
7. Liver function: Alanine transaminase(ALT), Aspartate aminotransferase(AST)< 1.5 times the upper limit of normal value (ULN), total bilirubin <1.0×ULN.
8. Renal function: serum creatinine <1×ULN.
9. Patients must sign informed consent and be willing and able to comply with the requirements of visits, treatment, laboratory tests and other research requirements stipulated in the research schedule.

Exclusion Criteria:

1. Histologically confirmed keratinizing squamous cell carcinoma (WHO I)
2. Suffered from other malignant tumors (except the cure of basal cell carcinoma or uterine cervical carcinoma in situ) previously.
3. Receiving radiotherapy or chemotherapy or targeted therapy previously
4. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the preparative chemotherapy on the fetus or infant.
5. Patients with significantly lower heart, liver, lung, kidney and bone marrow function.
6. Severe, uncontrolled medical conditions and infections.
7. At the same time using other test drugs or in other clinical trials.
8. Refusal or inability to sign informed consent to participate in the trial.
9. Emotional disturbance or mental illness, no civil capacity or limited capacity for civil conduct

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 366 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 2 years
  Defined from date of randomization to date of first documentation of progression or death due to any cause

SECONDARY OUTCOMES:
Overall survival | 2 years
  Defined from date of randomization to date of first documentation of death from any cause or censored at the date of the last follow-up.
Toxicities | 2 years
  Analysis of acute and late adverse events (AEs) are evaluated. Numbers of patients of treatment-related adverse events(acute toxicity) as assessed by CTCAE v5.0.Numbers of patients of late radiation toxicities were assessed using the Radiation Therapy Oncology Group and European Organization for Research and Treatment of Cancer late radiation morbidity scoring scheme.
change of quality of life | 1 year
  QoL scores were assessed for each scale by using the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire C30 (EORTCQLQ-C30) before induction chemotherapy, before radiotherapy, at the end of radiotherapy, at 3 months after radiotherapy, at 6 months after radiotherapy and 12 months after radiotherapy

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan Universtiy Shanghai Cancer Centre, Shanghai, Shanghai Municipality, China